CLINICAL TRIAL: NCT00883402
Title: Asymptomatic Carotid Surgery Trial-2 (ACST-2): an International Randomised Trial to Compare Carotid Endarterectomy With Carotid Artery Stenting to Prevent Stroke
Brief Title: Carotid Endarterectomy Versus Carotid Artery Stenting in Asymptomatic Patients
Acronym: ACST-2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: NHS Health Technology Assessment Programme (Other); BUPA Foundation (Other); British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ACST-2
Record Dates: First submitted 2009-04-15; First posted 2009-04-17 (Estimated); Last update posted 2024-12-09 (Actual); Status verified 2024-05

CONDITIONS: Carotid Stenosis
Keywords: Carotid stenosis; CEA; CAS; Stenting
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CEA (Active Comparator): Carotid endarterectomy
  Interventions: Procedure: CEA, CAS
- CAS (Active Comparator): Carotid Artery Stenting
  Interventions: Procedure: CEA, CAS

INTERVENTIONS:
Procedure: CEA, CAS — Carotid Artery Stenting (CAS) Carotid endarterectomy (CEA)

SUMMARY:
The trial randomise patients with asymptomatic carotid artery narrowing in whom prompt physical intervention is thought to be needed, but there there is still substantial uncertainty shared by patient and doctor about whether surgery or stenting is the more appropriate choice.

The study is looking at immediate risks (within one month)and at long term benefits

ELIGIBILITY:
Inclusion Criteria:

* Carotid artery stenosis detectable by duplex ultrasound, with no ipsilateral carotid territory symptoms(or none for some months) and no previous procedure done on it, which might well need procedural treatment now with CEA or CAS.
* Already started any appropriate medical treatment (eg, statin, aspirin etc), and already recovered from any necessary coronary procedures (eg, CABG)
* Patient seems fit and willing for follow-up in person (at 1 month) and by annual letter (for at least 5 years)
* Investigations show that both procedures (CEA and CAS) appear to be practicable and appropriate
* Some type of angiography (eg, MRA or CTA) has already been done that has shown that CEA and CAS would both be anatomically practicable.
* Doctor and patient both substantially uncertain about whether to treat with CEA or CAS, and the doctor sees no clear indication/contra-indication for either procedure

Exclusion Criteria:

* Small likelihood of worthwhile benefit (eg, very low risk of stroke because stenosis is very minor, or major co-morbidity or life-threatening disease, such as advanced cancer)
* Unsuitable for one or other procedure (eg, stenosis at carotid siphon that is inaccessible for CEA, or complex vasculature below the stenosis that would hinder CAS, or patient unfit for major surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3638 (Actual)
Dates: Start 2008-01; Primary Completion 2020-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To compare peri-procedural risks (MI, stroke and death) within the first month after the allocated CEA or CAS and long-term (up to 5 or more years) prevention of stroke, particularly disabling or fatal stroke, in subsequent years. | 10 years
  To compare peri-procedural risks (MI, stroke and death) within the first month after the allocated CEA or CAS and long-term (up to 5 or more years) prevention of stroke, particularly disabling or fatal stroke, in subsequent years.

SECONDARY OUTCOMES:
To identify types of patients to be identified in which one or other procedure is clearly preferable as well as economic evaluation; procedural costs and stroke-related healthcare costs and quality of life. | 10 years
  To identify types of patients to be identified in which one or other procedure is clearly preferable as well as economic evaluation; procedural costs and stroke-related healthcare costs and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Halliday, Principal Investigator — University of Oxford
Locations (125):
- University of Toledo Medical Centre, Toledo, Ohio, United States
- Medical University of Innsbruck, Innsbruck, Austria
- Belgium (6):
  - University Hospital Antwerp, Antwerp
  - University St Lucas, Brussels
  - Az St Blasius, Dendermonde
  - University Hospital Gent, Ghent
  - Centre Hospitalier Régional de la Citadelle, Liège
  - Centre Hospitalier De Mouscron, Mouscron
- Brazil (2):
  - HCFM Ribeirao Preto da Universidade de Sao Paulo, São Paulo
  - University of Sao Paulo, São Paulo
- Sveta Marina Hospital, Varna, Bulgaria
- Foothills Medical Centre, Calgary, Canada
- China (2):
  - China-Japan Friendship Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
- Croatia (2):
  - University Hospital Centre Zagreb, Zagreb
  - University Hospital of Merkur, Zagreb
- Czechia (5):
  - St Anne's University Hospital Brno, Brno
  - Hospital Ceské Budejovice, České Budějovice
  - Regional Hospital Liberec, Liberec
  - University Hospital Ostrava Poruba, Ostrava Poruba
  - Central Military Hospital, Prague
- Kasr Alaini University Hospital, Cairo, Egypt
- East Tallinn general Hospital, Tallinn, Estonia
- Henri Mondor University Hospital, Paris, France
- Germany (9):
  - University of Dresden 'Carl-Gustav-Carus', Dresden
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinik Jena, Jena
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - University of Leipzig, Leipzig
  - Universitätsmedizin Mannheim, Mannheim
  - Klinikum rechts der Isar derTechnischen Universität Muenchen, Munich
  - St Franziskus-Hospital Münster GmbH, Münster
  - Hegau-Bodensee-Klinikum, Singen
- Greece (3):
  - Democritus University of Thrace, Alexandroupoli
  - Dept. of Vascular Surgery, Attikon University Hospital, Athens
  - University Hospital of Larissa, Larissa
- Hungary (2):
  - Semmelweis Medical University, Budapest
  - Albert Szent-Györgyi Medical Centre, Szeged
- St. James' Hospital, Dublin, Ireland
- Rambam Hospital, Haifa, Israel
- Italy (32):
  - Cefalu Fondazione Istituto G.Giglio, Cefalù, PA
  - Azienda Ospedaliera S.G Moscati, Avellino
  - University of Bari, Bari
  - University of Bologna, Bologna
  - Policlinico Catania, Catania
  - Azienda Ospedaliero-Universitaria S.Anna, Ferrera
  - San Giovanni Di Dio, Florence
  - Opsedale Villa Scassi, Genoa
  - IRCCS San Martino, Genoa
  - Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico di Milano, Milan
  - IRCCS Policlinico San Donato, Milan
  - Istituto Auxologico Italiano, Milan
  - San Paolo Hospital, Milan
  - Mirano Hospital, Mirano
  - Nuovo Ospedale Civile Sant' Agostino Estense, Modena
  - Policlinico di Monza, Monza
  - Ospedale San Francesco di Nuoro, Nuoro
  - University of Palermo, Palermo
  - Foundation IRCCS Policlinico San Matteo, Pavia
  - Vascular Endovascular Unit of Perugia, Perugia
  - Santa Maria Hospital - Reggio, Raggio
  - Policlinico Universitario Campus Bio-medico di Roma, Roma
  - A.C.O. San Fillippo Neri, Rome
  - Fondazione Policlinico U. Agostino Gemeli IRCCS, Rome
  - San Camillo Forlanini, Rome
  - University La Sapienza, Rome
  - IRCCS Clinico Humanitas, Rozzano
  - Santa Maria alle Scotte, Siena
  - Ospedali Riuniti di Trieste, Trieste
  - Umberto I- ASO Mauriziano, Turin
  - Circolo University Hospital, Varese
  - San Giacomo Hospital, Veneto
- Sendai Medical Centre, Sendai, Japan
- National Scientific Centre of Surgery, Almaty, Kazakhstan
- Netherlands (3):
  - Rijnstate Hospital, Arnhem
  - MCL Leeuwarden, Leeuwarden
  - University Hospital Utrecht, Utrecht
- Rikshospitalet, Oslo, Norway
- Poland (6):
  - Poznan University of Medical Sciences, Poznan
  - Bielanski Hospital, Warsaw
  - Central Hospital Internal Aff., Warsaw
  - Mazovian Brodnowski Hospital, Warsaw
  - University of Warsaw/ Institute of Psychiatry, Warsaw
  - Regional Specialist Hospital (Wroclaw), Wroclaw
- Hospital Santa Marta, Lisbon, Portugal
- Russia (3):
  - Novosibirsk Research Institute of Circulation Pathology, Novosibirsk
  - Saint Petersburg Scientific Research Institute for Emergency Care, Saint Petersburg
  - V.A. Almazov National Medical Research Centre, Saint Petersburg
- Serbia (2):
  - Dedinje Cardiovascular Unit, Belgrade
  - Serbian Clinical Centre, Belgrade
- Institute of Medical Sciences, Ružomberok, Slovakia
- Slovenia (2):
  - Izola General Hospital, Izola
  - Teaching Hospital Maribor, Maribor
- Spain (3):
  - Hospital Clinic 1 Provinical de Barcelona, Barcelona
  - Guadalajara Hospital, Guadalajara
  - Hospital Universitari I Politecnic La Fe, Valencia
- Sweden (3):
  - Lasarettet Helsingborg, Helsingborg
  - Malmo University Hospital, Malmo
  - Sodersjukhuset, Stockholm
- Switzerland (2):
  - Cantonal Hospital Aarau, Aarau
  - University of Basel, Basel
- United Kingdom (24):
  - Southend University Hospital, Westcliff-on-Sea, Essex
  - East Kent Hospitals University NHS Foundation Trust, Canterbury, Kent
  - Walton Centre, Aintree
  - Cheltenham General Hospital, Cheltenham
  - Bishop Auckland Hospital, Durham
  - University Hospital of North Durham, Durham
  - Hull Royal Infirmary, Hull
  - St George's Hospital, London
  - The Royal London, London
  - Luton & Dunstable Hospital, Luton
  - Manchester Royal Infirmary, Manchester
  - Wythenshawe Hospital, Manchester
  - James Cook Hospital, Middlesbrough
  - Freeman Hospital, Newcastle
  - Royal Victoria Infirmary, Newcastle
  - Nottingham University Hospital, Nottingham
  - John Radcliffe Hospital, Oxford
  - Derriford Hospital, Plymouth
  - The Royal Preston Hospital, Preston
  - Royal Berkshire, Reading
  - Sheffield Vascular Institute, Sheffield
  - Sunderland Royal Hospital, Sunderland
  - Great Western Hospital, Swindon
  - North Cumbria University Hospital, Whitehaven

REFERENCES:
- [Background] Halliday A, Mansfield A, Marro J, Peto C, Peto R, Potter J, Thomas D; MRC Asymptomatic Carotid Surgery Trial (ACST) Collaborative Group. Prevention of disabling and fatal strokes by successful carotid endarterectomy in patients without recent neurological symptoms: randomised controlled trial. Lancet. 2004 May 8;363(9420):1491-502. doi: 10.1016/S0140-6736(04)16146-1. PMID 15135594
- See also: ACST-2 Website — http://www.acst-2.org